CLINICAL TRIAL: NCT03924349
Title: The Feasibility and Efficacy of ICG-coated Endoscopic Clip for Tumor Localization in Laparoscopic Colorectal Surgery
Brief Title: ICG-coated Endoscopic Clip for Tumor Localization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Dae Kyung Sohn, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NCC2019-0046
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective single center open label early phase clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG clip (Experimental): Three clips are fixed in three directions (120 degrees apart) at the distal of the lesion (just distal) before surgery
  Interventions: Device: ICG-coated clip

INTERVENTIONS:
Device: ICG-coated clip — Tumor localization using ICG-coated clip prior to surgery

SUMMARY:
The fluorescent clipping method involves endoscopic clipping a fluorescent clip into the colonic lesion site in advance of surgery, and observing the position of the fluorescence through the colonic wall by a light source of a certain wavelength band during surgery.

The purpose of this study is to evaluate the efficacy of the localization of colonic lesions using ICG coated endoscopic clip in laparoscopic colon surgery.

ELIGIBILITY:
Inclusion Criteria:

* Cases which are deemed necessary to mark the location of the colon lesion before surgery

Exclusion Criteria:

* Preoperative colonoscopy is not possible due to intestinal obstruction
* If the lesion is located in the rectal area and the lesion can be confirmed by digital rectal exam
* disagreement with the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Success rate of localization | through study completion, an average of 1 year
  The rate of Identifying ICG-coated clip during surgery

SECONDARY OUTCOMES:
loss rate of clips | through study completion, an average of 1 year
  The rate of detachment of clips before surgery
Number of Participants with Complication | through study completion, an average of 1 year
  Procedure-related complication

CONTACTS AND LOCATIONS:
Overall Officials: DAE KYUNG SOHN, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hyun JH, Kim SK, Kim KG, Kim HR, Lee HM, Park S, Kim SC, Choi Y, Sohn DK. A novel endoscopic fluorescent band ligation method for tumor localization. Surg Endosc. 2016 Oct;30(10):4659-63. doi: 10.1007/s00464-016-4785-1. Epub 2016 Feb 19. PMID 26895900
- [Result] Choi Y, Kim KG, Kim JK, Nam KW, Kim HH, Sohn DK. A novel endoscopic fluorescent clip for the localization of gastrointestinal tumors. Surg Endosc. 2011 Jul;25(7):2372-7. doi: 10.1007/s00464-010-1557-1. Epub 2011 Feb 7. PMID 21298528
- [Result] Hyun JH, Han KS, Kim BC, Hong CW, Oh JH, Park SC, Kim MJ, Sohn DK. Preoperative endoscopic clipping for rectal tumor localization in laparoscopic anterior resection. Minim Invasive Ther Allied Technol. 2019 Dec;28(6):326-331. doi: 10.1080/13645706.2018.1547765. Epub 2018 Dec 4. PMID 30513228
- [Result] Lee SJ, Sohn DK, Han KS, Kim BC, Hong CW, Park SC, Kim MJ, Park BK, Oh JH. Preoperative Tattooing Using Indocyanine Green in Laparoscopic Colorectal Surgery. Ann Coloproctol. 2018 Aug;34(4):206-211. doi: 10.3393/ac.2017.09.25. Epub 2018 Jul 26. PMID 30048996